CLINICAL TRIAL: NCT01017809
Title: Pilot Study Exploring the Efficacy of Prolonged Emend to Reduce Nausea and Vomiting During Treatment in a Phase II Study (NYU 03-67) of Oxaliplatin Combined With Continuous Infusion Topotecan for Patients With Previously Treated Ovarian Cancer
Brief Title: Prolonged Emend in a Study (NYU 03-67) of Oxaliplatin and Topotecan in Previously Treated Ovarian Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: NYU 03-67 reached accrual prior to this study opening.
Sponsor: NYU Langone Health (Other)
Responsible Party: Franco Muggia, MD, New York University Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NYU 08-851
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Ovarian Cancer
Keywords: ovarian; chemotherapy; nausea
MeSH Terms: conditions — Ovarian Neoplasms; Nausea | interventions — Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxali/Topotecan (Other): Patients enrolled to NYU 03-67 will be receiving Oxaliplatin 85 mg/m2 IV over 120 minutes on Day 1 and 15 Topotecan 0.4mg/m2/day CIV from D1 to 15 (in addition to the assigned intervention)
  Interventions: Drug: Aprepitant

INTERVENTIONS:
Drug: Aprepitant — Cycle 1, day 2 to 17: Emend 80mg once daily in the morning on days 2 through 17 Cycles 2-6 (optional extension arm): same Emend dosing
  Other Names: Emend

SUMMARY:
The investigators propose to totally abolish the emesis (vomiting) associated with the regimen of oxaliplatin + topotecan by adding a daily administration of aprepitant (Emend) for 17 days to the HT3 blocker routinely given on days 1 and 15.

DETAILED DESCRIPTION:
Patients enrolled in NCT0031361, NYU 03-67 (A Phase II study of Oxaliplatin combined with continuous infusion topotecan as chemotherapy for patients with previously treated ovarian cancer NCI #6317) will receive oxaliplatin 85mg/m2 as a 2-hr IV infusion on D1, 15 and topotecan 0.4mg/m2/day as a continuous infusion for 14 days beginning on D1 (D1-15) on a 4 week cycle.

On days 1 and 15 of the first cycle, patients will also receive IV ondansetron 32 mg and 10mg of dexamethasone. Emend 125 mg will be given on day 1; on days 2-17, patients will be given daily oral 80mg Emend without dexamethasone.

On cycles 2-6 patients opting to continue to receive Emend as above: Emend 125 mg will be given on day 1; on days 2-17, patients will be given daily oral 80mg Emend without dexamethasone.

Following cycle 1, Emend will be given in its conventional schedule (i.e., d 1-3, and d 15-17) unless after discussion with the Principal Investigator, the patient's request to receive drug as in cycle 1 is deemed desirable and safe to enter the optional extension arm.

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfilling the requirement for entering the study NYU 03-67 will be eligible to enter the supplementary protocol with Emend. Please see NCT0031361 for eligibility.

Exclusion Criteria:

* Patients not enrolled on NYU 03-67(NCT0031361).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
to determine whether daily administration of Emend will prevent emesis during cycle 1 in patients with previously treated ovarian cancer enrolled in NYU 03-67 (oxaliplatin combined with continuous infusion topotecan) | 28 days (1 cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Franco Muggia, MD, Principal Investigator — New York University Cancer Institute
Locations (1):
- NYU Clinical Cancer Center, New York, New York, United States